CLINICAL TRIAL: NCT00372008
Title: A Phase II Randomised, Two-Way Crossover Study to Compare the Steady State Pharmacokinetics of Testosterone Following Application of Different Testosterone Metered-Dose (MD) Lotion Doses in Hypogonadal Male Subjects
Brief Title: Pharmacokinetics of Testosterone Lotion in the Treatment of Hypogonadal Males
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acrux DDS Pty Ltd (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MTE05
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

INTERVENTIONS:
Drug: Testosterone

SUMMARY:
Testosterone replacement treatment is the most effective way of treating hypogonadism in men. Acrux has a proprietry testosterone replacement product - Testosterone-MD Lotion, and this study will evaluate the efficacy and safety of this product.

ELIGIBILITY:
Inclusion Criteria:

* Hypogonadal males between 18-70 years old with qualifying general medical health

Exclusion Criteria:

* Disqualifying concurrent conditions or allergy/sensitivity to testosterone replacement therapy

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic

SECONDARY OUTCOMES:
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Tina Soulis, PhD, Study Director — Acrux Ltd
Locations (7):
- United States (7):
  - Birmingham, Birmingham, Alabama
  - La Mesa, California
  - Torrance, California
  - New Britain, Connecticut
  - Ocala, Florida
  - Shreveport, Louisiana
  - San Antonio, Texas